CLINICAL TRIAL: NCT04737148
Title: The Analysis and Accuracy of Mortality Prediction Scores in Burn Patients Admitted to the Intensive Care Burn Unit (ICBU)
Brief Title: Analysis and Accuracy of Mortality Prediction Scores
Status: Completed | Type: Observational
Sponsor: Ministry of Health, Kuwait (Other Government)
Responsible Party: Principal Investigator, Zakariya Hassan, Assistant Registrar in plastic surgery, Ministry of Health, Kuwait
Other Study IDs: 14422
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Burns; Morality
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Mortality scores — Revised Baux, BOBI and FLAMES scores

SUMMARY:
Patients admitted to the ICU in a tertiary burn centre in Kuwait were analysed using multiple mortality prediction scores. The accuracy of these scores were compared to each other to ascertain which prediction modality provides the most accurate prognosis.

DETAILED DESCRIPTION:
The aim of this study is to determine the accuracy of three established scoring systems used for burn patients admitted to the intensive care unit and to determine the risk factors associated with poor outcomes.

A total of 211 patients with who were admitted to the ICBU in a tertiary care centre in Kuwait from January 2017 to December 2019 were analysed retrospectively. Data were collected using patient medical records. The FLAMES, BOBI and revised Baux scores were calculated, and the survivor and non-survivor scores of patients were analysed to determine the sensitivity, specificity and Area Under the Receiver Operating Characteristics (AUROC) of the different scoring modalities.

ELIGIBILITY:
Inclusion Criteria:

Pediatric burn patients with partial/full thickness burns>10% TBSA Adult patients with partial/full thickness burns >15% TBSA Patients with electric burns Patients iwth burns involving the voice Any patient with suspected inhalational injury Burn patients with significant comorbidities

Exclusion criteria:

Patients with incomplete data records

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to the ICBU between January 2017 to December 2019
Sampling Method: Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Area under curve of the 3 aforementioned mortality prediction scores | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- AlBabtain Centre for burns and plastic Surgery, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No